CLINICAL TRIAL: NCT02273960
Title: Open Label, Adaptive Design, Ascending, Multiple-Dose Study to Evaluate Safety and Efficacy of BMS-986004 in Adult Subjects With Primary Immune Thrombocytopenia (ITP)
Brief Title: Study to Evaluate Safety and Efficacy in Adult Subjects With ITP
Acronym: ITP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM140-103; 2014-001429-33 (EudraCT Number)
Record Dates: First submitted 2014-10-03; First posted 2014-10-24 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: BMS-986004 (Experimental): BMS-986004 solution intravenously (IV) as specified
  Interventions: Drug: BMS-986004 75 mg IV
- Arm B: BMS-986004 (Experimental): BMS-986004 solution intravenously as specified
  Interventions: Drug: BMS-986004 225 mg IV
- Arm C: BMS-986004 (Experimental): BMS-986004 solution intravenously as specified
  Interventions: Drug: BMS-986004 675 mg IV
- Arm D: BMS-986004 (Experimental): BMS-986004 solution intravenously as specified
  Interventions: Drug: BMS-986004 1500 mg IV

INTERVENTIONS:
Drug: BMS-986004 75 mg IV — BMS-986004 (75 mg) infusion (50 ml) administered in 120 minutes
  Arms: Arm A: BMS-986004
Drug: BMS-986004 225 mg IV — BMS-986004 (225 mg) infusion (100 ml) administered in 120 minutes
  Arms: Arm B: BMS-986004
Drug: BMS-986004 675 mg IV — BMS-986004 (675 mg) infusion (100 ml) administered in 120 minutes
  Arms: Arm C: BMS-986004
Drug: BMS-986004 1500 mg IV — BMS-986004 (1500 mg) infusion (100 ml) administered in 120 minutes
  Arms: Arm D: BMS-986004

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BMS-986004 when administered in subjects with ITP.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* ≥18 years old, diagnosed with persistent or chronic ITP

Exclusion Criteria:

* Secondary immune thrombocytopenia
* Drug induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (6):
  - Univ. Of Southern Calif. /Norris Comprehensive Cancer Center, Los Angeles, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Mass General Hospital, Boston, Massachusetts
  - Rutgers- Robert Wood Johnson Medical School, New Brunswick, New Jersey
- Australia (2):
  - Local Institution, Randwick, New South Wales
  - Local Institution, Brisbane, Queensland
- Hamilton Health Sciences/Mc Master Univ Med Ctre, Hamilton, Ontario, Canada
- Local Institution, Tbilisi, Georgia
- Local Institution, Chisinau, Moldova
- Poland (3):
  - Oddzial Kliniczny Hematologii i Profilaktyki Chorob Nowotworowych, Chorzów
  - Specjalistyczny Gabinet Lekarski Prof. dr hab. Krzysztof Giannopoulos, Lublin
  - Local Institution, Warsaw
- Russia (2):
  - Local Institution, Saint Petersburg
  - Local Institution, Smolensk
- United Kingdom (4):
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Glasgow, Lanarkshire
  - Local Institution, London

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bmsstudyconnect.com/us/en/home.html
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 participants were enrolled in the study and 26 participants entered the treatment period. Of the 20 who did not enter the treatment period, 19 did not meet study criteria and 1 experienced an adverse event.
Groups:
- BMS-986004 75mg IV: BMS-986004 dose level 75 mg
- BMS-986004 225mg IV: BMS-986004 dose level 225 mg
- BMS-986004 675 mg IV: BMS-986004 dose level 675 mg
- BM-986004 1500 mg IV: BMS-986004 dose level 1500 mg
Period: Short Term Period
Arm/Group | BMS-986004 75mg IV | BMS-986004 225mg IV | BMS-986004 675 mg IV | BM-986004 1500 mg IV
Started | 5 | 6 | 5 | 10
Completed (Completed = Entering Long Term Extension) | 0 | 0 | 1 | 4
Not Completed | 5 | 6 | 4 | 6
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — ST complete, not entering LTE | 4 | 6 | 4 | 5
Period: Long Term Extension
Arm/Group | BMS-986004 75mg IV | BMS-986004 225mg IV | BMS-986004 675 mg IV | BM-986004 1500 mg IV
Started | 0 | 0 | 1 | 4
Completed | 0 | 0 | 1 | 3
Not Completed | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- BMS 75 mg: BMS-986004 dose level 75 mg
- BMS 675mg: BMS-986004 dose level 675 mg
- BMS 1500mg: BMS-986004 dose level 1500 mg
- Total: Total of all reporting groups
Arm/Group | BMS 75 mg | BMS-986004 225mg IV | BMS 675mg | BMS 1500mg | Total
Number analyzed (Participants) | 5 | 6 | 5 | 10 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All treated participants
  Years | 52.8 (20.58) | 43.2 (16.33) | 34.2 (16.93) | 55.3 (16.09) | 48.0 (18.16)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Female | 2 | 2 | 4 | 4 | 12
    Male | 3 | 4 | 1 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 1 | 4 | 4 | 8 | 17
    Unknown or Not Reported | 4 | 2 | 1 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 1 | 1
    White | 4 | 5 | 5 | 7 | 21
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs): Short Term and Long Term
Description: The primary objective to establish safety was measured by the primary endpoints of AEs and SAEs for both Short term and Long term periods
Time Frame: Day 1 to Day 141 (Short term) and Day 1 to Day 398 (Long term)
Population: All participants who had received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Groups:
- BMS 225 mg: BMS-986004 dose level 225 mg
Arm/Group | BMS 75 mg | BMS 225 mg | BMS-986004 675 mg IV | BMS 1500mg
Number analyzed (Participants) | 5 | 6 | 5 | 10
Participants
  Number of participants with AEs | 1 | 5 | 5 | 9
  Number of participants with SAEs | 0 | 0 | 1 | 1

2. Primary Outcome: Number of ECG Abnormalities
Description: The primary objective to establish safety was measured by investigator identified Electrocardiogram Abnormalities for both Short term and Long term periods. ECG parameters included heart rate, PR interval, QRS interval, and QTcF interval (QT interval corrected for heart rate)
Time Frame: Day 1 to Day 141 (Short term) and Day 1 to Day 398 (Long term)
Population: All participants who had received at least 1 dose of study treatment
Measure: Number; unit: Events
Arm/Group | BMS 75 mg | BMS 225 mg | BMS-986004 675 mg IV | BMS 1500mg
Number analyzed (Participants) | 5 | 6 | 5 | 10
Events
  Screening | 1 | 3 | 2 | 3
  Day 1 | 1 | 2 | 2 | 3
  Day 71 | 0 | 2 | 0 | 0
  Day 72 | 1 | 0 | 1 | 1
  End of Treatment | 1 | 3 | 2 | 1
  LTE Day 1 | 0 | 0 | 0 | 2
  LTE Day 71 | 0 | 0 | 0 | 2
  End of LTE | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Laboratory Abnormalities of Safety Biomarkers: d-Dimer and Thrombin Anti-Thrombin (TAT)
Description: D-dimer and thrombin antithrombin (TAT) in plasma were quantified as measures of thromboembolism risk. D-dimer was evaluated by Enzyme linked immune sorbent assay (ELISA) method (D-dimer reference range 0-0.63 micrograms/milliliters fibrinogen equivalent units [mcg/ml FEU]). TAT reference range 0-4.1 ng/ml.
Time Frame: Day 1 to Day 141 (Short term) and Day 1 to Day 398 (Long Term)
Population: All participants who had received at least 1 dose of study treatment
Measure: Number; unit: Events
Arm/Group | BMS 75 mg | BMS 225 mg | BMS-986004 675 mg IV | BMS 1500mg
Number analyzed (Participants) | 5 | 6 | 5 | 10
Events
  # of events: d-Dimer, Normal | 56 | 81 | 60 | 106
  # of events: d-Dimer, High | 12 | 14 | 15 | 17
  # of events: TAT Complex, Normal | 52 | 71 | 46 | 112
  # of events: TAT Complex, High | 21 | 30 | 31 | 28

4. Secondary Outcome: Response Rate (RR) of BMS-986004: Short Term and Long Term
Description: Overall Response Rate (ORR) was defined as the proportion of participants who achieved a complete response (CR) or response (R). CR was defined as platelet count ≥ 100,000/mm3 and absence of bleeding. R was defined as platelet count ≥ 30,000/mm3 and at least 2-fold increase from the baseline count and absence of bleeding.
Time Frame: Day 1 to Day 141 (Short term) and Day 1 to Day 398 (Long term)
Population: All participants who had received at least 1 dose of study treatment
Measure: Number; unit: Proportion of participants
Arm/Group | BMS 75 mg | BMS 225 mg | BMS-986004 675 mg IV | BMS 1500mg
Number analyzed (Participants) | 5 | 6 | 5 | 10
Proportion of participants
  RR during ST | 0.2 | 0.3 | 0.4 | 0.4
  RR during LTE: number analyzed (Participants) | 0 | 0 | 1 | 4
  RR during LTE |  |  | 0 | 0

5. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of BMS-986004
Description: Pharmacokinetic parameter (Cmax) of BMS-986004, derived from serum concentration versus time. who have adequate PK profiles. On study Day 57, non-responders in each treatment group other than the 1500 mg group were dose escalated to the starting dose of the next higher treatment group.
Time Frame: Day 1 (0 hour [h], 2h, 24h, 72h, 168h), Day 15 (0h), Day 29 (0h), Day 43 (0h, 168h), Day 57 (0h, 2h), Day 71 (0h, 2h, 24h, 96h, 168h), Day 85 (0h, 336h, 672h, 1008h, 1344h)
Population: Evaluable PK population defined as participants with adequate PK profiles. The number of analyzed participants in each arm at specified time points represent the actual number of subjects evaluated after intra-participant dose escalation once the participant had completed the response phase of the study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BMS 75 mg | BMS 225 mg | BMS-986004 675 mg IV | BMS 1500mg
Number analyzed (Participants) | 2 | 6 | 6 | 13
ng/mL
  Cmax Day 1: number analyzed (Participants) | 2 | 6 | 4 | 9
  Cmax Day 1 | 19353.5 (6131.32) | 59478.8 (10021.04) | 177706.3 (37924.30) | 296561.9 (119530.86)
  Cmax Day 71: number analyzed (Participants) | 0 | 4 | 6 | 13
  Cmax Day 71 |  | 62469.8 (27336.64) | 186981.0 (22216.82) | 373588.9 (89833.77)

6. Secondary Outcome: Area Under the Concentration-time Curve in One Dosing Interval [AUC(TAU)] of BMS-986004
Description: Pharmacokinetics of BMS-986004 were derived from serum concentration versus time data. AUC(TAU) = Area under the concentration-time curve in one dosing interval. On study Day 57, non-responders in each treatment group other than the 1500 mg group were dose escalated to the starting dose of the next higher treatment group.
Time Frame: as for outcome 5
Population: Evaluable PK Population. The number of analyzed participants in each arm at specified time points represent the actual number of subjects evaluated after intra-participant dose escalation once the participant had completed the response phase of the study.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | BMS 75 mg | BMS 225 mg | BMS-986004 675 mg IV | BMS 1500mg
Number analyzed (Participants) | 2 | 6 | 6 | 13
h*ng/mL
  AUC(TAU) Day 1: number analyzed (Participants) | 2 | 6 | 4 | 9
  AUC(TAU) Day 1 | 915500 (196460) | 3445000 (708290) | 11440000 (3041300) | 18370000 (7351000)
  AUC(TAU) Day 71: number analyzed (Participants) | 0 | 4 | 6 | 13
  AUC(TAU) Day 71 |  | 4408000 (3313000) | 11460000 (2124900) | 26500000 (9366800)

7. Secondary Outcome: Trough Observed Serum Concentration (Ctrough) of BMS-986004
Description: Pharmacokinetics of BMS-986004 were derived from serum concentration versus time data. Ctrough = Trough observed serum concentration. On study Day 57, non-responders in each treatment group other than the 1500 mg group were dose escalated to the starting dose of the next higher treatment group.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BMS 75 mg | BMS 225 mg | BMS-986004 675 mg IV | BMS 1500mg
Number analyzed (Participants) | 5 | 6 | 6 | 14
ng/mL
  Ctrough, Day 15: number analyzed (Participants) | 5 | 6 | 5 | 10
  Ctrough, Day 15 | 978.0 (1080.82) | 2373.0 (1182.00) | 7556.4 (1952.53) | 15282.5 (9710.77)
  Ctrough, Day 29: number analyzed (Participants) | 5 | 6 | 5 | 10
  Ctrough, Day 29 | 1011.4 (999.13) | 3157.7 (1458.85) | 10236.0 (3737.42) | 21353.6 (14144.90)
  Ctrough, Day 43: number analyzed (Participants) | 5 | 6 | 5 | 9
  Ctrough, Day 43 | 1207.0 (852.88) | 3527.7 (1576.34) | 9416.2 (4410.57) | 19105.3 (14980.50)
  Ctrough, Day 57: number analyzed (Participants) | 0 | 4 | 6 | 14
  Ctrough, Day 57 |  | 25339.5 (49053.16) | 3360.5 (1082.75) | 20553.1 (19099.39)
  Ctrough, Day 71: number analyzed (Participants) | 0 | 4 | 6 | 13
  Ctrough, Day 71 |  | 3466.0 (3209.75) | 8347.7 (3215.32) | 25057.3 (18007.59)
  Ctrough, Day 85: number analyzed (Participants) | 0 | 4 | 6 | 13
  Ctrough, Day 85 |  | 4018.8 (4099.35) | 9075.7 (4268.76) | 24308.9 (19213.61)

8. Secondary Outcome: Total Body Clearance (CLT) of BMS-986004
Description: Pharmacokinetics of BMS-986004 were derived from serum concentration versus time data. On study Day 57, non-responders in each treatment group other than the 1500 mg group were dose escalated to the starting dose of the next higher treatment group.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/H
Arm/Group | BMS 75 mg | BMS 225 mg | BMS-986004 675 mg IV | BMS 1500mg
Number analyzed (Participants) | 2 | 6 | 6 | 13
L/H
  CLT Day 1: number analyzed (Participants) | 2 | 6 | 4 | 8
  CLT Day 1 | 0.0789 (0.01514) | 0.0618 (0.01617) | 0.0561 (0.01395) | 0.0860 (0.03037)
  CLT Day 71: number analyzed (Participants) | 0 | 4 | 6 | 13
  CLT Day 71 |  | 0.0716 (0.04106) | 0.0611 (0.01449) | 0.0628 (0.02061)

9. Secondary Outcome: AUC Accumulation Index (AI_AUC) of BMS-986004
Description: AUC accumulation index (AI_AUC) = ratio of AUC(TAU) at steady state to AUC(TAU) after the first dose of BMS-986004. On study Day 57, non-responders in each treatment group other than the 1500 mg group were dose escalated to the starting dose of the next higher treatment group.
Time Frame: as for outcome 5
Population: Evaluable PK Population. Only participants with adequate PK profiles were included in the summary statistics; "0" participants analyzed indicates "no data were available for that cohort for this Summary Statistic"
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | BMS 75 mg | BMS 225 mg | BMS-986004 675 mg IV | BMS 1500mg
Number analyzed (Participants) | 0 | 0 | 0 | 12
Ratio |  |  |  | 1.7996 (0.597881)

ADVERSE EVENTS:
Time Frame: All SAEs were collected that occurred during 21 day screening period, a 12 week treatment period (6 weeks of response Phase and 6 weeks of remission phase) and a 1 month follow up period. The collection of nonserious AE information began at initiation of study drug and up to follow up.
Arm/Group | BMS-986004 75mg IV | BMS-986004 225mg IV | BMS 675mg | BMS 1500mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 2/5 | 1/10
Other Adverse Events (participants affected / at risk) | 1/5 | 5/6 | 5/5 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986004 75mg IV (N=5) | BMS-986004 225mg IV (N=6) | BMS 675mg (N=5) | BMS 1500mg (N=10)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986004 75mg IV (N=5) | BMS-986004 225mg IV (N=6) | BMS 675mg (N=5) | BMS 1500mg (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 4
Feeling cold (General disorders) | 0 | 0 | 0 | 1
Infusion site bruising (General disorders) | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Allergy to animal (Immune system disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Phlebitis infective (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Heart sounds abnormal (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Neurosis (Psychiatric disorders) | 0 | 0 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Exercise lack of (Social circumstances) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT02273960/Prot_000.pdf
  • Statistical Analysis Plan (2015-01-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT02273960/SAP_001.pdf